CLINICAL TRIAL: NCT00152126
Title: Busulfan and Melphalan With Autologous Hematopoietic Stem Cell Support With Positively-Selected CD133+ Hematopoietic Cells for Children With High Risk Solid Tumors and Lymphomas
Brief Title: Chemotherapy With CD133+ Select Autologous Hematopoietic Stem Cells for Children With Solid Tumors and Lymphomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Miami (Other)
Responsible Party: Gregory Hale, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST133
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Neuroblastoma; Central Nervous System Tumors; Lymphomas; Wilms Tumor
Keywords: Autologous stem cell transplantation; CD133 cell selection; CliniMACS device; Tumor marker; Tumor purging
MeSH Terms: conditions — Neuroblastoma; Central Nervous System Neoplasms; Lymphoma; Wilms Tumor | interventions — Stem Cell Transplantation; Busulfan; Melphalan; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Stem Cell Transplantation; Drug: Busulfan, Melphalan

INTERVENTIONS:
Procedure: Stem Cell Transplantation — Autologous stem cell transplantation
Drug: Busulfan, Melphalan — Transplant recipients will receive high dose Busulfan and Melphalan followed by autologous CD133+ antigen specific hematopoietic stem cell infusion. The autologous graft product will be selected using the investigational CliniMACS device.
  Other Names: Autologous stem cell transplant; CD133+ antigen specific selection; Apheresis

SUMMARY:
Studies have provided evidence that residual microscopic malignant cells in autologous bone marrow or blood stem cell grafts can contribute to posttransplant relapse. Researchers are currently exploring different methods in an attempt to purify or "purge" the stem cell product to minimize the risk of tumor contamination.

The CD133+ antigen is a protein contained on or "expressed" on numerous cells in the human body including specific hematopoietic progenitor (blood forming) cells. However, this antigen is not expressed on certain cancer cells including neuroblastoma. A technique using the investigational CliniMACS cell sorting device has been developed in an effort to filter out only those stem cells that express this CD133+ antigen in order to infuse a hematopoietic stem cell product with no tumor contamination potential.

The primary objective of this study is to establish safety of treating patients with a high dose chemotherapy regimen of Busulfan and Melphalan followed by autologous CD133+ hematopoietic stem cell support. Transplants recipients are expected to achieve engraftment as defined by an absolute neutrophil count of greater than or equal to 500/mm3 for three consecutive days by day 42-post infusion. Thus, safety of the treatment plan will be evaluated in terms of failure to engraft by this specific time period.

DETAILED DESCRIPTION:
Secondary objectives for this protocol include the following:

* To describe CD133+ graft content post-selection and to describe the yield and purity of CD133+ content of the graft obtained.
* To describe the negative selection efficiency of this strategy by assessing the processed product for tumor specific markers, when applicable.
* To characterize the proliferation of clonal progeny of CD133+ cells.
* To characterize lymphocyte and hematopoietic reconstitution (including the kinetics of platelet engraftment) in these patients.
* To estimate one-year disease-free and overall survival in these transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

Eligibility will be determined separately for Part I and Part II of this study:

Part I ( Part I Eligibility criteria (eligibility for undergoing apheresis procedure)

* Age ≤ 25 years at initial diagnosis.
* Must have one of the following diagnoses:
* High risk neuroblastoma
* Metastatic or recurrent retinoblastoma
* High risk rain tumors
* Recurrent or refractory Hodgkin disease
* Recurrent or advanced stage Wilms tumor
* Recurrent or metastatic sarcomas
* Recurrent or refractory non-Hodgkin lymphoma
* Desmoplastic small round cell tumor.
* Lansky or Karnofsky Performance Score ≥ 70.
* Creatinine ≤ 2.0 mg/dl.
* Direct bilirubin ≤ 2.0 mg/dl.
* SGPT ≤ 2 x upper limit of normal
* HIV testing
* Negative pregnancy test
* Patients with significant prior radiation therapy to the liver will be excluded.

Part II eligibility criteria (criteria for transplantation of CD133 select stem cell product)

* Successfully completed Part I of protocol treatment plan and has the following available:
* Stored autologous bone marrow or peripheral blood stem cells (i.e. 2 x 106 unselected CD34+ cells/ kg PBSC or 1 x 106 CD34+ cells/ kg BM) for back up.
* Stored autologous bone marrow or peripheral blood stem cells (2 x 106 CD133+ cells/ kg PBSC or 2 x 106 CD133+ cells/ kg BM) for infusion.
* Forced vital capacity greater than or equal to 40% normal or pulse oximetry greater than or equal to 92% on room air.
* Lansky or Karnofsky Performance Score ≥ 70.
* Creatinine ≤ 2.0 mg/dl.
* Direct bilirubin ≤ 2.0 mg/dl.
* SGPT ≤ 2 x upper limit of normal
* Negative pregnancy test
* Patients with significant prior radiation therapy (in opinion of the PI) to the liver will be excluded.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2003-08; Primary Completion 2005-08 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety of the treatment plan using Busulfan and Melphalan followed by infusion of CD133+ selected hematopoietic cells in patients with high-risk malignancies. | August 2005

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hale, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org